CLINICAL TRIAL: NCT06038656
Title: Effects of Exercise and Acute and Chronic Galactooligosaccharide Supplementation on Inflammation and Iron Absorption in Female Athletes
Brief Title: Exercise and Galactooligosaccharide Supplementation on Inflammation and Iron Absorption (FexerGOS)
Acronym: FexerGOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North-West University, South Africa (Other)
Collaborators: Swiss Federal Institute of Technology (Other); King's College London (Other)
Responsible Party: Principal Investigator, Linda Malan, Associate Professor, North-West University, South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F_ExerGOS
Record Dates: First submitted 2023-08-31; First posted 2023-09-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Resistance Exercise
Keywords: Galacto-oligosaccharides; female athletes; iron absorption; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Participants will receive 10 g of GOS daily for 6 weeks. Fractional iron absorption will be determined pre- and post the 6-week intervention from 3 conditions: 1) after a period of rest; 2) three hours after an acute resistance exercise bout without GOS and 3) three hours after an acute resistance exercise bout, co-administered with 10 g GOS.
  Interventions: Dietary Supplement: Galactooligosaccharides (GOS)

INTERVENTIONS:
Dietary Supplement: Galactooligosaccharides (GOS) — 10 g of GOS provided as 14 g of powder will be consumed after mixing it in water or yoghurt.
  The absorption study test drinks administered during the 3 test conditions will be comprised as follows:
  Post rest period - 50 mg of iron as ferrous fumarate (Fefum) supplement, 6 mg 54Fe as Fefum and 300 ml of water with sucrose and lactose.
  Post exercise bout - 50 mg of iron as Fefum, 6 mg 58Fe as Fefum and 300 ml of water with sucrose and lactose.
  Post exercise bout co-administered with GOS - 50 mg of iron as Fefum, 6 mg 57Fe as Fefum and 300 ml of water with 10 g GOS.

SUMMARY:
Iron depletion is common in female athletes depending on the sports discipline. Endurance and resistance exercise can induce inflammation thereby reducing dietary iron absorption. Galacto-oligosaccharides (GOS) improved iron absorption in young healthy women and infants, and improved gut inflammation in iron-supplemented infants. A stable isotope study will be performed to investigate the effect exercise and acute and chronic GOS supplementation on inflammation and iron absorption in female athletes.

DETAILED DESCRIPTION:
Iron depletion is common in athletes, particularly in females, reaching prevalence rates up to 70% depending on the sports discipline. As iron is essential for energy production and oxygen transport, a deficiency can impair performance, especially in endurance athletes. Iron deficiency in athletes may be caused by inadequate intake, but reduced iron absorption and increased losses also seem to play a role. Both endurance and resistance exercise at a high intensity, can induce inflammation resulting in a hepcidin response via interleukin-6 (IL-6) regulation. Hepcidin is the master regulator of systemic iron homeostasis, and a recent study in adult males showed that vigorous exercise decreases dietary iron absorption associated with increases in IL-6 and hepcidin. Iron losses induced by exercise have been attributed to several factors, including gastrointestinal bleeding associated with endothelial damage, haematuria, haemolysis, and increased sweating. Galacto-oligosaccharides (GOS) have been shown to acutely enhance iron absorption in young, healthy women. In Kenyan infants with a high infectious disease burden, chronic GOS administration improved iron absorption and mitigated the negative effects of iron supplementation on gut inflammation, likely mediated by its bifidogenic effect. Whether GOS has the potential of improving iron absorption has not been studied in athletes.

The study aims are to determine 1) the effects of a bout of resistance exercise at 70% 1 repetition maximum (RM) on inflammation, hepcidin and iron absorption in female team athletes; and 2) the effect of acute and chronic GOS supplementation on iron absorption in response to the exercise bout.

The trial will entail two series of three iron absorption conditions separated by six weeks of GOS supplementation (10 g/day). The study participants will be 22 female athletes recruited from the North-West University and Potchefstroom area, South Africa. At baseline, the first series of three iron absorption studies will be conducted, all measuring iron absorption from a supplement administered with labelled ferrous fumarate in the following conditions: 1) after a period of rest; 2) three hours after an acute resistance exercise bout; and 3) three hours after an acute resistance exercise bout, co-administered with GOS. Following this, participants will consume GOS daily for 6 weeks, followed by an identical series of iron absorption studies. Markers of systemic and gut inflammation, hepcidin, microflora composition and iron status indicators before and after the GOS intervention will be determined. In addition, erythrocyte iron incorporation will be determined after both series of isotope studies. Furthermore, the kinetics of isotope appearance, inflammatory markers, and hepcidin for 24 hours during each of the six iron absorption studies will be investigated.

The primary hypotheses are that fractional iron absorption from a supplemental dose of ferrous fumarate will be: 1) lower three hours post exercise than post resting period; 2) higher with co-administration of GOS than without, both before and after six-week GOS intervention; and 3) higher after six-week intervention with GOS compared to baseline.

The secondary hypotheses are: 1) acute exercise bout will result in increased inflammatory and hepcidin response before and after intervention with GOS but the intervention may mediate these two responses; 2) chronic GOS intervention will increase relative abundance of Bifidobacterium spp, reduce gut inflammation and improve gut integrity and gut health; 3) chronic GOS intervention will improve iron status.

ELIGIBILITY:
Inclusion Criteria:

1. Female athlete.
2. Train at least 6 hours per week at moderate to high intensity.
3. Having low to moderate iron stores.
4. Willingness to consume the study supplement GOS during the intervention period.
5. Willingness not to consume daily nutritional supplements containing >20 mg iron and/or pre- or probiotics (excluding food and beverages containing live cultures such as yoghurt, raw milk and cheese) during the study.
6. Willingness to not take any iron-containing supplements two days before and during the iron absorption study days or vitamin C on the iron absorption study days.

Exclusion Criteria:

1. Haemoglobin <11 g/dl.
2. Treated or self-reported chronic disease, malabsorptive or gastrointestinal disorders (e.g. irritable bowel syndrome, functional bloating).
3. Pregnancy or lactation.
4. Subjects who cannot be expected to comply with the study protocol.
5. Difficulty drawing blood due to poor quality veins.
6. Individuals that have a fear of needles or suffer from vaso-vagal episodes when exposed to blood.
7. Participants who plan to start or stop the use of contraceptives before or during study period.
8. Participants who are lactose intolerant.
9. Participants who donated blood in the past 4 months or plan to donate during the study period.
10. Participants who use chronic anti-inflammatory medication such as corticosteroids or non-steroidal anti-inflammatory medication (NSAIDS).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
a. Fractional iron absorption (%) | Visit 8 (day 29) and 15 (day 92).
  Fractional iron absorption will be measured at rest and after an exercise bout.
b. Fractional iron absorption (%) | Visit 8 (day 29) and 15 (day 92).
  Fractional iron absorption will be measured after an exercise bout with and without co-administration of GOS.
c. Fractional iron absorption (%) | Visit 8 (day 29) and 15 (day 92).
  Fractional iron absorption will be measured at rest and after an exercise bout before and after a 6-week intervention with GOS.

SECONDARY OUTCOMES:
Interleukin 6 (pg/mL) | Visits 2 (day 1), 3 (day 2), 4 (day 8), 5 (day 9), 6 (day 15), 7 (day 16), 9 (day 64), 10 (day 65), 11 (day 71), 12 (day 72), 13 (day 78) and 14 (day 79)
  Interleukin 6 (IL-6) will be measured over 24 hours after rest and after exercise as a marker of exercise-induced inflammation.
C-reactive protein (mg/L) | Visits 2 (day 1), 4 (day 8), 6 (day 15), 9 (day 64), 11 (day 71) and 13 (day 78).
  C-reactive protein (CRP) will be measured in plasma to detect the presence of acute inflammation.
Alpha-1-acid glycoprotein (g/L) | Visits 2 (day 1), 4 (day 8), 6 (day 15), 9 (day 64), 11 (day 71) and 13 (day 78).
  Alpha-1-acid glycoprotein (AGP) will be measured in plasma to determine the presence of chronic inflammation.
Hepcidin (ng/mL) | Visits 2 (day 1), 3 (day 2), 4 (day 8), 5 (day 9), 6 (day 15), 7 (day 16), 9 (day 64), 10 (day 65), 11 (day 71), 12 (day 72), 13 (day 78) and 14 (day 79)
  Hepcidin, a major regulator of iron absorption and influenced by exercise-induced inflammation, will be measured in plasma over 24 hours.
Lipid mediators (pg/µL ) | Visits 2 (day 1), 3 (day 2), 4 (day 8), 5 (day 9), 6 (day 15), 7 (day 16), 9 (day 64), 10 (day 65), 11 (day 71), 12 (day 72), 13 (day 78) and 14 (day 79)
  The following lipid mediators will be measured over 24 hours in plasma in response to exercise-induced inflammation:17-hydroxydocosahexaenoicacid (17-HDHA); 5-, 8-, 9-, 11-, 12-, 15 and 18- hydroxyeicosapentaenoicacid (HEPE); 5-, 8-, 11-, 12- and 15-hydroxyeicosatetraenoicacid (HETE); prostaglandin (PG) E2 and D2, and resolvin (Rv) D1 and E1).
Erythropoietin (mIU/mL) | Visits 2 (day 1), 4 (day 8), 6 (day 15), 9 (day 64), 11 (day 71) and 13 (day 78).
  Plasma erythropoietin, a marker of erythropoiesis, will be measured before and after period of rest and exercise.
Serum iron isotope (%) | Visits 2 (day 1), 3 (day 2), 4 (day 8), 5 (day 9), 6 (day 15), 7 (day 16), 9 (day 64), 10 (day 65), 11 (day 71), 12 (day 72), 13 (day 78) and 14 (day 79).
  Kinetics of serum iron isotope appearance during a period of rest and post-exercise, before and after intervention with GOS, and with and without co-administration of GOS.
Gut microbial composition | Visit 8 (day 29) and 15 (day 92).
  Gut microbiota profile will be assessed at baseline and endpoint.
Faecal short chain fatty acids (µmol/g) | Visit 8 (day 29) and 15 (day 92).
  Concentration of short chain fatty acids - acetate, propionate, isobutyrate, butyrate, formate, isovalerate will be measured in faecal samples before and after the 6-week intervention with GOS.
Faecal pH | Visit 8 (day 29) and 15 (day 92).
  Faecal pH will be measured at baseline and endpoint to determine a response to the GOS intervention.
Faecal calprotectin (µg/g) | Visit 8 (day 29) and 15 (day 92).
  Faecal calprotectin will be measured at baseline and endpoint as a marker of gut inflammation.
Faecal zonulin (ng/mL) | Visit 8 (day 29) and 15 (day 92).
  Faecal zonulin will be measured at baseline and endpoint as a marker of the integrity of the intestinal mucosal barrier.
Intestinal fatty acid-binding protein (pg/mL) | Screening, Visits 4 (day 8), 8 (day 29), 9 (day 64), 11 (day 71) and 15 (day 92).
  Intestinal fatty acid-binding protein (I-FABP), a marker of intestinal damage, will be measured in plasma at baseline and endpoint.
Haemoglobin (g/dL) | Screening,Visit 8 (day 29), 9 (day 64) and 15 (day 92).
  Haemoglobin will be measured in whole blood to determine presence of anaemia and for calculation of fractional iron absorption.
Ferritin (µg/L) | Screening, Visits 2 (day 1) and 9 (day 64).
  Ferritin will be measured in plasma to determine the presence of iron deficiency.
Soluble transferrin receptor (mg/L) | Screening, Visits 2 (day 1) and 9 (day 64).
  Soluble transferrin receptor (sTfR) will be measured in plasma to determine the presence of iron deficiency.
Retinol-binding protein 4 (µmol/L) | Screening, Visits 2 (day 1) and 9 (day 64).
  Retinol-binding protein 4 (RBP4) will be measured in plasma as a marker of vitamin A status.
Thyroglobulin (µg/L) | Screening, Visits 2 (day 1) and 9 (day 64).
  Thyroglobulin will be measured in plasma as a marker of iodine status.
Fibroblast growth factor 21 (pg/mL) | Screening,Visits 2 (day 1) and 9 (day 64).
  Fibroblast growth factor 21 (FGF-21) will be measured in plasma as a marker of environmental enteric dysfunction (EED).
Insulin-like growth factor 1 | Screening, Visits 2 (day 1) and 9 (day 64).
  Insulin-like growth factor 1 (IGF-1) will be measured in plasma as on of the markers of environmental enteric dysfunction.
Dietary intake | Screening, Visit 8 (day 29) and 15 (day 92).
  Dietary intake will be captured using a quantified food frequency questionnaire.
Method comparison in the measurement of RBP4 (µmol/L) | Screening
  Two methods will be compared in the measurement of RBP4 (µmol/L).
Method comparison in the measurement of Ferritin (µg/L) | Screening
  Two methods will be compared in the measurement of Ferritin (µg/L).
Method comparison in the measurement of sTfR (mg/L) | Screening
  Two methods will be compared in the measurement of sTfR (mg/L).
Method comparison in the measurement of CRP (mg/L) | Screening
  Two methods will be compared in the measurement of CRP (mg/L).
Method comparison in the measurement of AGP (g/L) | Screening
  Two methods will be compared in the measurement of AGP (g/L).
Method comparison in the measurement of I-FABP (pg/mL) | Screening
  Two methods will be compared in the measurement of I-FABP (pg/mL).
Method comparison in the measurement of Thyroglobulin (µg/L) | Screening
  Two methods will be compared in the measurement of Thyroglobulin (µg/L).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, Principal Investigator — ETH Zurich; Jesslee du Plessis, Principal Investigator — North-West University
Locations (1):
- Este Vorster Research Facility, Potchefstroom, North West, South Africa

IPD SHARING:
Plan to Share IPD: No